CLINICAL TRIAL: NCT02373410
Title: Effect of the Height of the Operating Table During Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: I-2014-6010
Record Dates: First submitted 2014-11-27; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2014-09

CONDITIONS: Anesthesia, Spinal [E03.155.086.331]; Operating Tables [E07.325.662]
MeSH Terms: interventions — Body Piercing; Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Umbilicus (Experimental): The height of the operating table which set at the needle insertion point, is the level of umbilicus of the anesthesiologist in a standing posture.
  Interventions: Procedure: Umbilicus; Drug: Umbilicus Bupivacaine
- Lowest rib margin (Active Comparator): The height of the operating table which set at the needle insertion point, is the level of lowest rib margin of the anesthesiologist in a standing posture.
  Interventions: Procedure: Lowest rib margin; Drug: Lowest rib margin Bupivacaine
- Xiphoid (Active Comparator): The height of the operating table which set at the needle insertion point, is the level of xiphoid of the anesthesiologist in a standing posture.
  Interventions: Procedure: Xiphoid; Drug: Xiphoid Bupivacaine
- Nipple (Active Comparator): The height of the operating table which set at the needle insertion point, is the level of nipple of the anesthesiologist in a standing posture.
  Interventions: Procedure: Nipple; Drug: Nipple Bupivacaine

INTERVENTIONS:
Procedure: Umbilicus — Depending on the height of the operating table, the insertion angle of the spinal needles would be vary. The investigators intend to find the optimal angle and the height of the table to provide that.
  The height of the operating table which set at the needle insertion point of anesthetists; the level of umbilicus
  Arms: Umbilicus
Procedure: Lowest rib margin — The height of the operating table which set at the needle insertion point of anesthetists; the level of lowest rib margin
  Arms: Lowest rib margin
Procedure: Xiphoid — The height of the operating table which set at the needle insertion point of anesthetists; the level of xiphoid
  Arms: Xiphoid
Procedure: Nipple — The height of the operating table which set at the needle insertion point of anesthetists; the level of nipple
  Arms: Nipple
Drug: Umbilicus Bupivacaine — If freely flowing of CSF is detected, appropriate dose of MARCAINE was injected in all interventional groups.
  Other Names: Bupivacaine
  Arms: Umbilicus
Drug: Lowest rib margin Bupivacaine — If freely flowing of CSF is detected, appropriate dose of MARCAINE was injected in all interventional groups.
  Other Names: Bupivacaine
  Arms: Lowest rib margin
Drug: Xiphoid Bupivacaine — If freely flowing of CSF is detected, appropriate dose of MARCAINE was injected in all interventional groups.
  Other Names: Bupivacaine
  Arms: Xiphoid
Drug: Nipple Bupivacaine — If freely flowing of CSF is detected, appropriate dose of MARCAINE was injected in all interventional groups.
  Other Names: Bupivacaine
  Arms: Nipple

SUMMARY:
The purpose of this study is to analyze the accuracy of needle insertion and the discomfort during different ergonomic conditions faced by anesthesiologists during spinal anesthesia. In particular,the investigators intend to compare the angles between the patients' back and the inserted spinal needle in the coronal plane at different operating table heights.

DETAILED DESCRIPTION:
Sixty patients will be recruited undergoing elective surgery under spinal anesthesia. The patients will be randomly allocated to one of four groups: Group U, L, X, and N. These acronyms indicate the heights of the operating table which set at the needle insertion point of anesthetists, namely the level of umbilicus, lowest rib margin, xiphoid process, and nipple in a standing posture. The angle between the patient's skin and the spinal needle will be measured by the protractor in the coronal and sagittal plane. The anesthesiologists will be asked to record the subjective general discomfort graded by Numeric Rating Scale. And the degree of neck, lower back, knee, and elbow flexion of the anesthesiologists will be measured by taking pictures during procedure.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective surgery under spinal anesthesia

Exclusion Criteria:

* body mass index (BMI)>30
* history of spine operation or severe anatomical abnormalities of spine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The angle between the patient's skin and the spinal needle | during procedure

SECONDARY OUTCOMES:
anesthesiologist's subjective discomfort | during procedure
the degree of anesthesiologist's joint flexion | during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jinhee Kim, MD,PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyeonggido, South Korea

REFERENCES:
- [Background] Lee HC, Yun MJ, Hwang JW, Na HS, Kim DH, Park JY. Higher operating tables provide better laryngeal views for tracheal intubation. Br J Anaesth. 2014 Apr;112(4):749-55. doi: 10.1093/bja/aet428. Epub 2013 Dec 18. PMID 24355831
- [Background] Ajmal M, Power S, Smith T, Shorten GD. An ergonomic task analysis of spinal anaesthesia. Eur J Anaesthesiol. 2009 Dec;26(12):1037-42. doi: 10.1097/EJA.0b013e3283317dc9. PMID 19707143